



# STATISTICAL ANALYSIS PLAN

# SPD422, Anagrelide Hydrochloride PHASE 1

A Phase 1, Open-label, Single-sequence, Non-randomized, Crossover, Drug-Drug Interaction Study to Evaluate the Effect of Omeprazole on the Pharmacokinetics of SPD422 (anagrelide hydrochloride) in Healthy Adult Subjects

**PROTOCOL IDENTIFIER: SPD422-113** 

**Study Sponsor(s)**: Shire

300 Shire Way, Lexington, MA 02421 USA

Author:

Protocol: 2018 OCT 04 Original

SAP Version #: 1.0

SAP Date: 2019 MAY 08

Status: Final

Shire 

Shire Statistical Analysis Plan v1.0 Protocol Number: SPD422-113

08 May 2019

# REVISION HISTORY

| Version | Issue Date | Summary of Changes |
|---------|------------|------------------------|
| 1.0 | 08MAY2019 | Original final version |

# TABLE OF CONTENTS

| REV | ISION HISTORY | 2 |
|------|--------------------------------------------------|----|
| TABI | LE OF CONTENTS | 3 |
| ABBI | REVIATIONS | 6 |
| 1. | INTRODUCTION | 8 |
| 2. | OBJECTIVES, ESTIMANDS, AND ENDPOINTS | 8 |
| 2.1 | 1 Objectives | 8 |
| | 2.1.1 Primary Objective | 8 |
| | 2.1.2 Secondary Objective | 8 |
| 2.2 | 2 Endpoints | 8 |
| | 2.2.1 Primary Endpoints | 8 |
| | 2.2.2 Secondary Endpoints | 8 |
| 3. | STUDY DESIGN | 8 |
| 3.1 | l General Description | 8 |
| 3.2 | | |
| 3.3 | Blinding | 9 |
| 3.4 | 4 Sample Size and Power Considerations | 9 |
| 4. | STATISTICAL ANALYSIS SETS | 10 |
| 4.1 | 1 Enrolled Set | 10 |
| 4.2 | 2 Safety Set | 10 |
| 4.3 | 3 Pharmacokinetic Set | 10 |
| 5. | STUDY SUBJECTS | 11 |
| 5.1 | 1 Disposition of Subjects | 11 |
| 5.2 | 2 Demographic and Other Baseline Characteristics | 11 |
| 5.3 | 3 Medical History | 12 |
| 5.4 | 4 Prior Medications | |
| 5.5 | | |
| 5.6 | Exposure to Investigational Product | |
| 5.7 | 7 Measurements of Treatment Compliance | |
| 5.8 | 8 Protocol Deviations | 13 |

| 6. | EFFICACY ANALYSES | 13 |
|---|---|---|
| 7. | SAFETY ANALYSIS | 14 |
| 7. | .1 Adverse Events | 14 |
| 7. | .2 Clinical Laboratory Data | 15 |
| 7. | .3 Vital Signs | 18 |
| 7. | .4 Electrocardiogram (ECG) | 18 |
| 7. | .5 Other Safety Data | 19 |
| 8. | PHARMACOKINETIC ANALYSIS | 19 |
| 8. | .1 Drug Concentration | 19 |
| 8. | .2 Handling Below Limit of Quantitation Values | 20 |
| 8. | .3 Pharmacokinetic Parameters | 20 |
| 8. | .4 Statistical Analysis of Pharmacokinetic Data | 20 |
| 9. | OTHER ANALYSES | 21 |
| 10. | INTERIM ANALYSIS/ DATA MONITORING COMMITTEE | 23 |
| 11. | DATA HANDLING CONVENTIONS | 23 |
| 1 | 1.1 General Data Reporting Conventions | 23 |
| 1 | 1.2 Definition of Baseline | 23 |
| 1 | 1.3 Repeated or Unscheduled Assessments of Safety Parameters | 23 |
| 1 | 1.4 Handling of Missing, Unused, and Spurious Data | 23 |
| | 11.4.1 Missing Date Information for Prior or Concomitant Medications | |
| | (Therapies/Procedures) | 23 |
| | 11.4.1.1 Incomplete Start Date | 24 |
| | 11.4.1.2 Incomplete Stop Date | 24 |
| | 11.4.2 Missing Date Information for Adverse Events | 25 |
| | 11.4.2.1 Incomplete Start Date | 25 |
| | 11.4.2.2 Incomplete Stop Date | 25 |
| | 11.4.3 Missing Severity Assessment for Adverse Events | |
| | 11.4.4 Missing Relationship to Investigational Product for Adverse Events | 26 |
| | 11.4.5 Character Values of Clinical Laboratory Variables | 26 |

| Snire<br>Statisti | cal Analysis Plan v1.0 | Page 5 01 31 |
|-------------------|-------------------------------------------|--------------|
| | ol Number: SPD422-113 | 08 May 2019 |
| 12. | ANALYSIS SOFTWARE | 26 |
| 13. | CHANGES TO ANALYSIS SPECIFIED IN PROTOCOL | 26 |
| 14. | REFERENCES | 27 |
| 15. | APPENDICES | 28 |
| 15. | 1 Schedule of Activities | 28 |

Shire 

Statistical Analysis Plan v1.0 Protocol Number: SPD422-113

otocol Number: SPD422-113 08 May 2019

#### **ABBREVIATIONS**

AE adverse event

ANOVA analysis of variance AUC area under the curve

 $AUC_{0-\infty}$  area under the curve extrapolated to infinity

 $AUC_{0-t}$  area under the curve from time 0 to the last time point of sample

collection

AUC<sub>0-tau</sub> area under the curve from time 0 to the end of the dosing interval (24

hours post dose)

BLQ below limit of quantitation

BMI body mass index
CI confidence interval
CL/F total body clearance
Cmax maximum concentration

C<sub>min</sub> minimum concentration observed over the dosing interval C<sub>trough</sub> Plasma concentration observed at the end of a dosing interval

CV coefficient of variation ECG electrocardiogram

eCRF electronic case report form EM extensive metabolizer

IM/PM intermediate metabolizers/poor metabolizer

LLOQ lower limit of quantification

MedDRA Medical Dictionary for Regulatory Activities

MR metabolite ratio

PCI potentially clinically important

PK pharmacokinetic(s)
PT preferred term
Q1 25th Percentile
Q3 75th Percentile
QD once daily

QTcB QT interval corrected for heart rate using Bazett's formula QTcF QT interval corrected for heart rate using Fridericia's formula

SAP statistical analysis plan SD standard deviation SOC system organ class t½ terminal half-life

TEAE treatment-emergent adverse event

TFL tables, figures, and listings

t<sub>max</sub> time of maximum observed concentration sampled during a dosing

interval

Shire 

Statistical Analysis Plan v1.0 Protocol Number: SPD422-113

ocol Number: SPD422-113 08 May 2019

V<sub>z</sub>/F volume of distribution associated with the terminal slope following

extravascular administration

WHO World Health Organization

#### 1. INTRODUCTION

This statistical analysis plan (SAP) provides a technical and detailed elaboration of the statistical analyses of pharmacokinetic (PK) and safety data described in the original study protocol dated 04 Oct 2018. Specifications for tables, figures, and listings (TFLs) are contained in a separate document (SPD422-113 TFL Shells).

#### 2. OBJECTIVES, ESTIMANDS, AND ENDPOINTS

# 2.1 Objectives

# 2.1.1 Primary Objective

The primary objective of this study is to assess the effect of a CYP1A2 inducer (omeprazole) on the PK of an agrelide when administered concurrently.

# 2.1.2 Secondary Objective

The secondary objective of this study is to assess the safety and tolerability of anagrelide, omeprazole, and co-administered anagrelide plus omeprazole.

# 2.2 Endpoints

# 2.2.1 Primary Endpoints

The primary endpoints will be maximum concentration ( $C_{max}$ ) and area under the curve from time 0 to the last time point of sample collection (AUC<sub>0-t</sub>) and area under the curve extrapolated to infinity (AUC<sub>0-∞</sub>) of an agrelide and 3-hydroxyanagrelide compared between an agrelide administered alone and an agrelide administered after ome prazole 40 mg once daily (QD) for 7 days.

# 2.2.2 Secondary Endpoints

Safety and tolerability will be assessed throughout the study by routine recording of electrocardiograms (ECGs), vital signs, safety laboratory assessments, and adverse events (AEs).

#### 3. STUDY DESIGN

#### 3.1 General Description

This is a Phase 1, open-label, single-sequence, non-randomized, multiple-dose, crossover PK study to assess the effect of a CYP1A2 inducer (omeprazole 40 mg QD) on the PK of anagrelide (1 mg) when administered concurrently in healthy subjects. Up to 35 healthy

male and female subjects, aged 18 to 45 years will be screened to ensure enrollment and completion of 20 subjects. Subjects who discontinue from the study will not be replaced. The study design is shown in the study schema in Figure 1.

Figure 1: Study Design Flow Chart



- SPD422 will be administered under fasting conditions on Days 1 and 8
- Omeprazole will be administered prior to breakfast on Days 2-7 and under fasting conditions on Day 8
- PK assessments for anagrelide on Day 1 and Day 8, and for omeprazole on Day 8

#### 3.2 Randomization

Not applicable.

# 3.3 Blinding

Not applicable.

#### 3.4 Sample Size and Power Considerations

Up to 35 healthy male and female subjects, aged 18 to 45 years will be screened to ensure enrollment and completion of 20 subjects. Subjects who discontinue will not be replaced.

08 May 2019

Sample size estimation is to achieve a desired precision of the effect of interest, targeting the width of the 90% confidence interval (CI).

From a previous crossover study (SPD422-110), the within-subject coefficient variation (CV) in anagrelide log-transformed AUC was estimated to be 0.132. Allowing for a slightly larger within-subject CV of 0.15, a sample size of 11 subjects is required to estimate the mean difference between anagrelide + omeprazole and anagrelide alone in the log-transformed AUC with an error margin of at most  $\pm 0.2231$  at 90% confidence with a probability of 90%. Thus, if the true geometric mean treatment ratio is 0.6, the lower and upper 90% confidence bounds will be estimated to be within 0.48 and 0.75 (exp[ln(0.6) - 0.2231] and exp[ln(0.6) + 0.2231]) with 90% probability. Therefore, with an overall sample size of 20 subjects, anticipated 13 to 14 CYP2C19 extensive metabolizer (EM) subjects and 6 to 7 CYP2C19 intermediate/poor metabolizer (IM/PM) subjects, this statistical power will be met for the overall population and the CYP2C19 EM population. The confidence bounds for the smaller population of CYP2C19 IM/PM subjects will be slightly wider.

#### 4. STATISTICAL ANALYSIS SETS

#### 4.1 Enrolled Set

The Enrolled Set consists of all subjects for whom an enrollment number has been assigned. Usually, these are the subjects who meet the study inclusion/exclusion criteria and sign the informed consent form.

#### 4.2 Safety Set

The Safety Set consists of all subjects who have taken at least 1 dose of investigational product (anagrelide or omeprazole) and have at least 1 post-dose safety assessment.

#### 4.3 Pharmacokinetic Set

The PK Set consists of subjects who receive at least 1 dose of investigational product (anagrelide or omeprazole) and have at least 1 measurable post-dose plasma concentration. Each subject's data (eg, dosing records, AEs, sample collection records, etc.) will be reviewed for inclusion/exclusion from the descriptive statistics and statistical analysis on a case-by-case basis at the discretion of the Pharmacokineticist.

#### 5. STUDY SUBJECTS

## 5.1 Disposition of Subjects

The number of subjects who were included in each defined analysis set (Enrolled, Safety, and PK) will be summarized overall.

The number and percentage of subjects who completed the study or prematurely discontinued will be presented overall, along with primary reasons for discontinuation, as recorded on the study completion/early termination page of the electronic case report form (eCRF). All enrolled subjects who prematurely discontinued the study will be listed in the subject disposition listing along with reasons for discontinuation.

Subject disposition summary and listings will be based on the Enrolled Set.

# 5.2 Demographic and Other Baseline Characteristics

Descriptive summaries of demographic and baseline characteristics will be generated for the Safety Set and the PK Set.

The observed omeprazole AUC<sub>0-tau</sub> will be used to define the CYP2C19 metabolizer status of subjects, with AUC<sub>0-tau</sub> <5,200 ng•h/mL (<15  $\mu$ mol/L) classified as CYP2C19 EM and AUC<sub>0-tau</sub>  $\geq$ 5,200 ng•h/mL ( $\geq$ 15  $\mu$ mol/L) classified as CYP2C19 IM/PM. The summaries of demographic and baseline characteristics for the PK Set will be presented by the CYP2C19 metabolizer status (EMs and IMs/PMs) and overall.

The following demographic and baseline characteristics will be summarized in the following order in the tables: age (years), sex, ethnicity, race, weight (kg), height (cm), and body mass index (BMI, kg/m<sup>2</sup>).

Continuous variables, such as age, weight, height, and BMI will be summarized using descriptive statistics including number of subjects, mean, standard deviation (SD), median, minimum, and maximum. Categorical variables such as sex, ethnicity and race will be summarized by reporting the number and percentage of subjects in each category. All summarized values will be taken from the latest available assessments at the Screening Visit.

Demographic and baseline characteristics will be listed for the Safety Set.

08 May 2019

#### 5.3 Medical History

Medical history will be collected at the Screening visit and will be coded using Medical Dictionary for Regulatory Activities (MedDRA) Version 21.1. A listing will be provided using the Safety Set.

Medical history will be summarized by system organ class (SOC) and preferred term (PT) for the Safety Set.

#### 5.4 Prior Medications

Prior medications will be coded using the World Health Organization (WHO) Drug Dictionary Enhanced Version dated 01 September 2018.

Prior medication is defined as any medication with the start date prior to the date of first dose of investigational product.

Prior medication usage will be summarized by the number and proportion of subjects receiving each medication by PT and overall for the Safety Set. Multiple medication usage by a subject in the same category will be counted only once.

All prior medications will be listed for the Safety Set.

#### 5.5 Concomitant Medications

Concomitant medications will be coded using the WHO Drug Dictionary Enhanced Version dated 01 September 2018.

Concomitant medication is defined as any medication with a start date prior to the date of the first dose of investigational product and continuing after the first dose of investigational product or with a start date between the dates of the first and last doses of investigational product, inclusive. Any medication with a start date after the date of the last dose of investigational product will not be considered a concomitant medication.

Concomitant medication usage will be summarized by the number and proportion of subjects receiving each medication by PT, by treatment group and overall, for the Safety Set. Multiple medication usage by a subject in the same category will be counted only once. Concomitant medications will be assigned to the treatment(s) with which they are concomitant. A medication is concomitant with a treatment if the subject received that medication any time between the time when that treatment was received and when the next treatment was received, or in the case of the last treatment, until the end of the

08 May 2019

follow-up period. Therefore, a medication may be concomitant with more than one treatment.

All concomitant medications will be listed for the Safety Set.

# 5.6 Exposure to Investigational Product

Exposure to investigational product for the Safety Set will be summarized in terms of treatment duration, which is calculated as the number of days from the date of first dose of investigational product taken to the date of the last dose of investigational product taken, inclusively. Descriptive statistics (number of subjects, mean, standard deviation, minimum, median, and maximum) will be presented to describe the exposure to investigational product.

A listing will be created by subject number and visit giving the date and time of dose administration for the Safety Set.

# 5.7 Measurements of Treatment Compliance

This is a study in which the investigational products will be administered from Day 1 to Day 8 at the study site only (in-house confinement treatment period). All compliance related data will be included in the exposure data listing. No separate treatment compliance summary or data listing will be provided.

#### 5.8 Protocol Deviations

Protocol deviations will be recorded by the site separately from the clinical database. Protocol deviations will be classified as major or minor per the agreed protocol deviation management plan. The Shire study team will review the protocol deviations and their classification throughout the study and before database lock.

Decisions of the review will include categorization of major and minor protocol deviations.

Confirmed major and minor protocol deviations will be documented in the protocol deviation tracker for the study. Major/minor protocol deviations will be summarized by category for the Safety Set. Major/minor protocol deviations will be listed for the Enrolled Set.

#### 6. EFFICACY ANALYSES

Not applicable.

#### 7. SAFETY ANALYSIS

The safety analysis will be performed using the Safety Set. Safety parameters include AEs, clinical laboratory results, vital signs, and ECG results. For each safety parameter, the last value collected prior to dosing on Day 1 will be used as baseline for all analyses of that safety parameter.

#### 7.1 Adverse Events

Adverse events will be coded using MedDRA Version 21.1.

An AE (classified by PT) will be considered a treatment-emergent AE (TEAE) if it starts on or after dosing on Day 1, or if it starts before dosing on Day 1 but increases in severity on or after dosing on Day 1 through the end of the study. If more than 1 AE with the same PT is reported before dosing on Day 1, then the AE with the greatest severity will be used as the benchmark for comparison to the AEs occurring after dosing on Day 1 under the PT.

Treatment most recently taken when the AE occurred will be used for the summaries:

- Any AE that started (or increased in severity) on or after the administration of anagrelide on Day 1, but before the administration of omeprazole on Day 2 will be assigned to anagrelide alone;
- Any AE that started (or increased in severity) on or after the administration of omeprazole on Day 2, but before the administration of anagrelide on Day 8 will be assigned to omeprazole alone;
- Any AE that started (or increased in severity) on or after the administration of anagrelide on Day 8 will be assigned to anagrelide with omeprazole.

An overall summary of the number of subjects with TEAEs as well as the number of events will be presented by treatment group, including the number and percentage of subjects with any TEAEs, serious TEAEs, TEAEs related to investigational product, serious TEAEs related to investigational product, TEAEs leading to discontinuation of investigational product, serious TEAEs leading to discontinuation of investigational product, TEAEs leading to discontinuation from study, serious TEAEs leading to discontinuation from study, severe TEAEs, TEAEs leading to hospitalization, and TEAEs leading to death.

08 May 2019

The number and percentage of subjects reporting TEAEs, as well as the number of events, in each treatment group and overall will be tabulated by SOC and PT, and by SOC, PT, and maximum severity. The TEAEs considered related to investigational product will also be summarized by SOC and PT. If more than 1 AE occurs with the same PT, after the same treatment for the same subject, then the subject will be counted only once for that treatment group and PT using the most severe and most related occurrence for the summarization by severity and by relationship to investigational product. Summaries by SOC and PT will present SOC sorted alphabetically and PT within SOC by descending incidence.

The TEAEs and related TEAEs will be summarized by PT by descending frequency. Serious TEAEs, TEAEs leading to discontinuation of investigational product and serious TEAEs leading to death, will be summarized by SOC, PT, and treatment group.

## 7.2 Clinical Laboratory Data

Descriptive statistics for clinical laboratory values (in SI units) and changes from baseline at each assessment time point as well as shift tables from baseline to each visit for quantitative variables will be presented by treatment group for the following clinical laboratory parameters:

**Hematology** Hemoglobin, hematocrit, red blood cells, platelet count, white blood cell

count – total and differential, total neutrophils (absolute), eosinophils (absolute), monocytes (absolute), basophils (absolute) and lymphocytes

(absolute).

**Biochemistry** Sodium, potassium, glucose, blood urea nitrogen, creatinine, calcium,

chloride, phosphorus, total protein, total CO2 (bicarbonate), albumin,

aspartate transaminase, alanine transaminase, gamma glutamyl transferase, alkaline phosphatase, total bilirubin, and uric acid.

**Urinalysis** pH, glucose, protein, blood, ketones, bilirubin, nitrites, leukocyte

esterase, and specific gravity.

Clinical laboratory test values are potentially clinically important (PCI) if they meet either the low or high PCI criteria listed in Table 1. The number and percentage of subjects with post-baseline PCI values will be tabulated overall. The percentages will be calculated relative to the number of subjects with available baseline values and at least 1 post-baseline assessment. The numerator is the total number of subjects with at least


1 post-baseline PCI value. A supportive listing of subjects with post-baseline PCI values will be provided including the subject number, baseline, and post-baseline values.

Table 1: Criteria for Potentially Clinically Important Laboratory Tests

| Parameter | Classification | Criteria: SI Units (Conventional Units) |
|---|---|---|
| Hematology | • | |
| | LOW and DECDEASE | <100 g/L (10g/dL) AND |
| Hematology Hemoglobin Hematocrit Red blood cells count Platelet count White blood cell count Neutrophils Eosinophils Monocytes Basophils Lymphocytes Biochemistry Sodium Potassium | LOW and DECREASE | Decrease of $\geq$ 20 g/L (2.0 g/dL) from baseline value |
| | HIGH | >200 g/L (20g/dL) |
| | LOW and DECREASE | ≤0.6 × LLN AND |
| Hematocrit | LOW and DECKEASE | Decrease of ≥0.06 L/L (6.0%) from baseline value |
| | HIGH | >1.3 × ULN |
| Pad blood calls count | LOW | $<3 \times 10^{12}/L$ |
| Red blood cells could | HIGH | $>7.5 \times 10^{12}/L$ |
| Distalat assumt | LOW | $<0.6 \times LLN OR < 100 \times 10^{9}/L (100 \times 10^{3}/\mu L)$ |
| Flatelet Coulit | HIGH | $>1.5 \times ULN OR > 500 \times 10^9/L (500 \times 10^3/\mu L)$ |
| White blood call count | LOW | $<0.5 \times LLN OR < 3.0 \times 10^{9}/L (3 \times 10^{3}/\mu L)$ |
| White blood cell count Neutrophils Eosinophils Monocytes Basophils Lymphocytes | HIGH | $>2 \times ULN OR > 16.0 \times 10^{9}/L (16 \times 10^{3}/\mu L)$ |
| Nautranhila | LOW | $<1.5 \times 10^9/L (1.5 \times 10^3/\mu L) OR < 40\%$ |
| Neutrophiis | HIGH | $>6.2 \times 10^9/L (6.2 \times 10^3/\mu L) OR > 70 \%$ |
| Eosinophils | HIGH | $>0.5 \times 10^9$ /L $(0.5 \times 10^3$ / $\mu$ L) OR $> 10.0$ % |
| Monocytes | HIGH | $>1.1 \times 10^9$ /L $(1.1 \times 10^3$ / $\mu$ L) OR $>11 \%$ |
| Basophils | HIGH | $>0.2 \times 10^9$ /L $(0.2 \times 10^3/\mu$ L) OR $> 2\%$ |
| Lymphagytag | LOW | $<0.8 \times 10^9$ /L $(0.8 \times 10^3$ / $\mu$ L) OR $< 22 \%$ |
| Lymphocytes | HIGH | $> 4.0 \times 10^9 / L (4.0 \times 10^3 / \mu L) OR > 44 \%$ |
| Biochemistry | | |
| Cadina | LOW | >5 mmol/L (5 mEq/L) below LLN |
| Soulum | HIGH | >5 mmol/L (5 mEq/L) above ULN |
| | | Below LLN AND |
| | LOW and DECREASE | Decrease of >0.5 mmol/L (0.5 mEq/L) from |
| Neutrophils Eosinophils Monocytes Basophils Lymphocytes Biochemistry Sodium | | baseline value |
| rotassium | | Above ULN AND |
| | HIGH and INCREASE | Increase of $> 0.5 \text{ mmol/L} (0.5 \text{ mEq/L}) \text{ from}$ |
| | | baseline value |
| Glucose (facting) | LOW | ≤4.2 mmol/L |
| Glucose (lasting) | HIGH | ≥6.7 mmol/L |
| Blood urea nitrogen | HIGH | >1.5 × ULN |
| Creatinine | HIGH and INCREASE | >150 µmol/L AND |
| Creatinine | IIIOII and INCKEASE | Increase > 30% from baseline value |
| | | Below LLN AND |
| Calcium | LOW and DECREASE | Decrease of ≥0.25 mmol/L (1.0 mg/dL) from |
| | | baseline value |

08 May 2019

| HIGH and INCREASE HIGH and INCREASE Increase of ≥ 0.25 mmol/L (1.0 mg/dL) from baseline value | Parameter | Classification | Criteria: SI Units (Conventional Units) |
|---|---|---|---|
| Baseline value Baseline value Phosphorus LOW Phosphorus Phosphorus Phosphorus LOW Phosphorus | | | Above ULN AND |
| Phosphorus | | HIGH and INCREASE | Increase of $\geq$ 0.25 mmol/L (1.0 mg/dL) from |
| Phosphorus HIGH >0.162 mmol/L (0.5 mg/dL) above ULN Total protein LOW and DECREASE Below LLN AND Decrease of ≥0 g/L (2.0 g/dL) from baseline value Albumin HIGH and INCREASE Above ULN AND Increase of ≥10 g/L (1.0 g/dL) from baseline value Albumin HIGH and INCREASE Below LLN AND Decrease of ≥10 g/L (1.0 g/dL) from baseline value Aspartate transaminase HIGH >2 × ULN Alanine transaminase HIGH >2 × ULN Gamma glutamyl transferase HIGH >1.5 × ULN Alkaline phosphatase HIGH >1.5 × ULN Uric acid (with normal diet) LOW and DECREASE Below LLN AND Decrease of >0.119 mmol/L (2.0 mg/dL) from baseline value Decrease of >0.119 mmol/L (2.0 mg/dL) from baseline value Triiodothyronine LOW <0.922 mmol/L | | | baseline value |
| Total protein | Dhaanhama | LOW | >0.162 mmol/L (0.5 mg/dL) below LLN |
| Total protein Company Decrease of ≥20 g/L (2.0 g/dL) from baseline value | Pnospnorus | HIGH | >0.162 mmol/L (0.5 mg/dL) above ULN |
| Decrease of ≥20 g/L (2.0 g/dL) from baseline value | | LOW and DECREASE | Below LLN AND |
| HIGH and INCREASE Above ULN AND Increase of ≥20 g/L (2.0 g/dL) from baseline value Below LLN AND Decrease of ≥10 g/L (1.0 g/dL) from baseline value Above ULN AND Increase of ≥0.119 mmol/L (2.0 mg/dL) from baseline value Above ULN AND Increase of ≥0.119 mmol/L (2.0 | Total protain | LOW and DECKEASE | Decrease of ≥20 g/L (2.0 g/dL) from baseline value |
| Increase of ≥20 g/L (2.0 g/dL) from baseline value Below LLN AND Decrease of ≥10 g/L (1.0 g/dL) from baseline value Above ULN AND Increase of ≥0.0 g/dL Above ULN AND Decrease of ≥0.0 g/dL Above ULN AND Decrease of >0.0 g/dL Above ULN AND Decrease of >0.0 g/dL Above ULN AND Increase of ≥0.0 g/dL Above ULN AND Increase of ≥0.0 g/dL Above ULN AND Increase of >0.0 g/dL Above ULN AND Incr | Total protein | HICH and INCDEASE | Above ULN AND |
| Albumin Decrease of ≥10 g/L (1.0 g/dL) from baseline value Albumin HIGH and INCREASE Decrease of ≥10 g/L (1.0 g/dL) from baseline value Aspartate transaminase HIGH >2 × ULN Alanine transaminase HIGH >2 × ULN Gamma glutamyl transferase HIGH >1.5 × ULN Alkaline phosphatase HIGH >1.5 × ULN Total bilirubin HIGH >1.5 × ULN Uric acid (with normal diet) LOW and DECREASE Below LLN AND Decrease of >0.119 mmol/L (2.0 mg/dL) from baseline value Decrease of >0.119 mmol/L (2.0 mg/dL) from baseline value Triiodothyronine LOW <0.922 nmol/L | | HIGH ally INCREASE | Increase of ≥20 g/L (2.0 g/dL) from baseline value |
| Albumin Decrease of ≥10 g/L (1.0 g/dL) from baseline value Aspartate transaminase HIGH and INCREASE Above ULN AND Increase of ≥10 g/L (1.0 g/dL) from baseline value Aspartate transaminase HIGH >2 × ULN Alanine transaminase HIGH >2 × ULN Gamma glutamyl transferase HIGH >1.5 × ULN Alkaline phosphatase HIGH >1.5 × ULN Total bilirubin HIGH >1.5 × ULN Uric acid (with normal diet) Below LLN AND Decrease of >0.119 mmol/L (2.0 mg/dL) from baseline value 2.922 nmol/L Thyroide trimulating hormone LOW <57.92 nmol/L | | LOW and DECREASE | Below LLN AND |
| Aspartate transaminase Aspartate transaminase Alanine transaminase Alanine transaminase Alanine transaminase Alanine transaminase Alanine transaminase HIGH Alanine transaminase HIGH Alanine transaminase HIGH Alanine phosphatase Alkaline phosphatase Alkaline phosphatase HIGH Total bilirubin HIGH Alanine phosphatase Alkaline phosphatase HIGH Alanine phosphatase Alkaline phosphatase HIGH Alanine phosphatase Alkaline phosphatase HIGH Alanine phosphatase Alkaline phosphatase HIGH Alanine phosphatase Alkaline phosphatase Alkaline phosphatase HIGH Alanine phosphatase Alkaline phosphatase Alkaline phosphatase HIGH Alanine phosphatase Alkaline Alkaline A | Alhumin | LOW and DECKEASE | Decrease of ≥10 g/L (1.0 g/dL) from baseline value |
| Aspartate transaminase Alanine transaminase Alanine transaminase HIGH Alanine transaminase HIGH Alanine transaminase HIGH Alanine transaminase HIGH Alanine transaminase HIGH Alanine phosphatase HIGH Alkaline phosphatase HIGH | Albuillii | HIGH and INCREASE | Above ULN AND |
| Alanine transaminase HIGH >2 × ULN | | THOH and INCREASE | Increase of ≥10 g/L (1.0 g/dL) from baseline value |
| Gamma glutamyl transferase HIGH >1.5 × ULN Alkaline phosphatase HIGH >1.5 × ULN Total bilirubin HIGH >1.5 × ULN Uric acid (with normal diet) LOW and DECREASE Below LLN AND Decrease of >0.119 mmol/L (2.0 mg/dL) from baseline value Triiodothyronine LOW <0.922 nmol/L | Aspartate transaminase | HIGH | >2 × ULN |
| transferase HIGH >1.5 × ULN Alkaline phosphatase HIGH >1.5 × ULN Total bilirubin HIGH >1.5 × ULN Uric acid (with normal diet) LOW and DECREASE Below LLN AND Decrease of >0.119 mmol/L (2.0 mg/dL) from baseline value Triiodothyronine LOW <0.922 nmol/L | Alanine transaminase | HIGH | >2 × ULN |
| transferase Alkaline phosphatase HIGH 7 total bilirubin HIGH Vic acid (with normal diet) HOW and DECREASE Below LLN AND Decrease of >0.119 mmol/L (2.0 mg/dL) from baseline value 1 | Gamma glutamyl | нісн | >1.5 × III.N |
| Total bilirubin HIGH >1.5 × ULN Uric acid (with normal diet) LOW and DECREASE Below LLN AND Decrease of >0.119 mmol/L (2.0 mg/dL) from baseline value Triiodothyronine LOW <0.922 nmol/L | transferase | IIIOII | >1.5 ^ OLIV |
| Uric acid (with normal diet)LOW and DECREASEBelow LLN AND Decrease of $>0.119 \text{ mmol/L}$ ( $2.0 \text{ mg/dL}$ ) from baseline valueTriiodothyronineLOW $<0.922 \text{ nmol/L}$ ThyroxineLOW $<57.92 \text{ nmol/L}$ Thyroid stimulating hormoneLOW $<57.92 \text{ nmol/L}$ Uric acid (with normal diet)LOW $<0.5 \mu \text{U/L}$ Uric acid (with normal diet)HIGH and INCREASEAbove ULN AND Increase of $<0.119 \text{ mmol/L}$ ( $<0.0 \text{ mg/dL}$ ) from baseline valueUrinalysisGlucoseHIGH $<0.0 \text{ mg/dL}$ ProteinHIGH $<0.0 \text{ mg/dL}$ BloodHIGH $<0.0 \text{ mg/dL}$ HIGH $<0.0 \text{ mg/dL}$ HIGH $<0.0 \text{ mg/dL}$ HIGH $<0.0 \text{ mg/dL}$ ProteinHIGH $<0.0 \text{ mg/dL}$ HIGH $<0.0 \text{ mg/dL}$ | Alkaline phosphatase | HIGH | >1.5 × ULN |
| Uric acid (with normal diet)LOW and DECREASEDecrease of $>0.119 \text{ mmol/L}$ ( $2.0 \text{ mg/dL}$ ) from baseline valueTriiodothyronineLOW $<0.922 \text{ nmol/L}$ ThyroxineLOW $<57.92 \text{ nmol/L}$ Thyroid stimulating hormoneLOW $<0.5 \mu \text{U/L}$ HIGH $>1.00 \text{U/L}$ Uric acid (with normal diet)HIGH and INCREASEAbove ULN AND Increase of $>0.119 \text{ mmol/L}$ ( $2.0 \text{ mg/dL}$ ) from baseline valueUrinalysisGlucoseHIGH $\ge 1+$ ProteinHIGH $\ge 2+$ BloodHIGH $\ge 2+$ KetonesHIGH $\ge 2+$ BilirubinHIGHPositiveNitritesHIGHPositive | Total bilirubin | HIGH | >1.5 × ULN |
| $\begin{array}{c ccccccccccccccccccccccccccccccccccc$ | Uric acid (with normal | | Below LLN AND |
| Triiodothyronine LOW <0.922 nmol/L HIGH >2.765 nmol/L Thyroxine LOW <57.92 nmol/L HIGH >140.28 nmol/L Thyroid stimulating hormone HIGH >5.0 μU/L Uric acid (with normal diet) HIGH and INCREASE Above ULN AND Increase of >0.119 mmol/L (2.0 mg/dL) from baseline value Urinalysis Glucose HIGH ≥1+ Protein HIGH ≥2+ Blood HIGH ≥2+ Ketones HIGH ≥2+ Ketones HIGH ≥2+ Ketones HIGH ≥2+ Blirubin HIGH Positive Nitrites HIGH Positive | , | LOW and DECREASE | Decrease of >0.119 mmol/L (2.0 mg/dL) from |
| $ \begin{array}{ c c c }\hline Triiodothyronine & HIGH & >2.765 \text{ nmol/L} \\ \hline Thyroxine & LOW & <57.92 \text{ nmol/L} \\ \hline HIGH & >140.28 \text{ nmol/L} \\ \hline Thyroid stimulating & LOW & <0.5 \mu\text{U/L} \\ \hline HIGH & >5.0 \mu\text{U/L} \\ \hline Uric acid (with normal diet) & HIGH and INCREASE & Above ULN AND & Increase of >0.119 mmol/L (2.0 mg/dL) from baseline value \\ \hline \textbf{Urinalysis} & & \\ \hline Glucose & HIGH & \geq 1+ & Protein & HIGH & \geq 2+ & Blood & HIGH & \geq 2+ & Ketones & HIGH & \geq 2+ & Bilirubin & HIGH & \geq 2+ & Bilirubin & HIGH & Positive & $ | uict) | | baseline value |
| $ \begin{array}{c ccccccccccccccccccccccccccccccccccc$ | Trijodothyronine | LOW | |
| Thyroxine $HIGH$ >140.28 nmol/L Thyroid stimulating hormone $HIGH$ <0.5 $\mu$ U/L Uric acid (with normal diet) $HIGH$ and INCREASE $HIGH$ = 21+ Protein $HIGH$ = 21+ Protein $HIGH$ = 22+ Blood $HIGH$ = 22+ Ketones $HIGH$ = 22+ Bilirubin $HIGH$ Positive Nitrites $HIGH$ Positive | Tinodothyronine | HIGH | >2.765 nmol/L |
| Thyroid stimulating hormone $IOW = 140.28 \text{ nmol/L}$ Thyroid stimulating hormone $IOW = 140.28 \text{ nmol/L}$ Uric acid (with normal diet) $IOW = 140.28 \text{ nmol/L}$ Uric acid (with normal diet) $IOW = 140.28 \text{ nmol/L}$ HIGH and INCREASE $IOW = 140.28 \text{ nmol/L}$ Above ULN AND Increase of >0.119 mmol/L (2.0 mg/dL) from baseline value Urinalysis Glucose $IOW = 140.28 \text{ nmol/L}$ HIGH $IOW = 140.28 \text{ nmol/L}$ Above ULN AND Increase of >0.119 mmol/L (2.0 mg/dL) from baseline value $IOW = 140.28 \text{ nmol/L}$ Above ULN AND Increase of >0.119 mmol/L (2.0 mg/dL) from baseline value $IOW = 140.28 \text{ nmol/L}$ Above ULN AND Increase of >0.119 mmol/L (2.0 mg/dL) from baseline value $IOW = 140.28 \text{ nmol/L}$ Above ULN AND Increase of >0.119 mmol/L (2.0 mg/dL) from baseline value $IOW = 140.28 \text{ nmol/L}$ Above ULN AND Increase of >0.119 mmol/L (2.0 mg/dL) from baseline value $IOW = 140.28 \text{ nmol/L}$ Above ULN AND Increase of >0.119 mmol/L (2.0 mg/dL) from baseline value $IOW = 140.28 \text{ nmol/L}$ Above ULN AND Increase of >0.119 mmol/L (2.0 mg/dL) from baseline value $IOW = 140.28 \text{ nmol/L}$ Above ULN AND Increase of >0.119 mmol/L (2.0 mg/dL) from baseline value $IOW = 140.28 \text{ nmol/L}$ Above ULN AND Increase of >0.119 mmol/L (2.0 mg/dL) from baseline value $IOW = 140.28 \text{ nmol/L}$ Above ULN AND Increase of >0.119 mmol/L (2.0 mg/dL) from baseline value $IOW = 140.28 \text{ nmol/L}$ $IOW $ | Thuravina | LOW | <57.92 nmol/L |
| hormoneHIGH>5.0 μU/LUric acid (with normal diet)HIGH and INCREASEAbove ULN AND Increase of >0.119 mmol/L (2.0 mg/dL) from baseline valueUrinalysisGlucoseHIGH $\geq 1+$ ProteinHIGH $\geq 2+$ BloodHIGH $\geq 2+$ KetonesHIGH $\geq 2+$ BilirubinHIGHPositiveNitritesHIGHPositive | Thyroxine | HIGH | >140.28 nmol/L |
| Uric acid (with normal diet) HIGH and INCREASE Above ULN AND Increase of >0.119 mmol/L (2.0 mg/dL) from baseline value Urinalysis Structure Glucose HIGH ≥1+ Protein HIGH ≥2+ Blood HIGH ≥2+ Ketones HIGH ≥2+ Bilirubin HIGH Positive Nitrites HIGH Positive | Thyroid stimulating | LOW | <0.5 μU/L |
| Uric acid (with normal diet) HIGH and INCREASE Increase of >0.119 mmol/L (2.0 mg/dL) from baseline value Urinalysis Glucose HIGH ≥1+ Protein HIGH ≥2+ Blood HIGH ≥2+ Ketones HIGH ≥2+ Bilirubin HIGH Positive Nitrites HIGH Positive | hormone | HIGH | >5.0 µU/L |
| diet) HIGH and INCREASE Increase of >0.119 mmol/L (2.0 mg/dL) from baseline value Urinalysis Glucose HIGH $\geq 1+$ Protein HIGH $\geq 2+$ Blood HIGH $\geq 2+$ Ketones HIGH $\geq 2+$ Bilirubin HIGH Positive Nitrites HIGH Positive | Urio goid (with normal | | Above ULN AND |
| baseline valueUrinalysisGlucoseHIGH $\geq 1+$ ProteinHIGH $\geq 2+$ BloodHIGH $\geq 2+$ KetonesHIGH $\geq 2+$ BilirubinHIGHPositiveNitritesHIGHPositive | ` | HIGH and INCREASE | Increase of >0.119 mmol/L (2.0 mg/dL) from |
| | uici) | | baseline value |
| ProteinHIGH $\geq 2+$ BloodHIGH $\geq 2+$ KetonesHIGH $\geq 2+$ BilirubinHIGHPositiveNitritesHIGHPositive | Urinalysis | | |
| BloodHIGH $\geq 2+$ KetonesHIGH $\geq 2+$ BilirubinHIGHPositiveNitritesHIGHPositive | Glucose | HIGH | ≥1+ |
| Ketones HIGH ≥2+ Bilirubin HIGH Positive Nitrites HIGH Positive | Protein | HIGH | ≥2+ |
| Bilirubin HIGH Positive Nitrites HIGH Positive | Blood | HIGH | ≥2+ |
| Nitrites HIGH Positive | Ketones | HIGH | ≥2+ |
| | Bilirubin | HIGH | Positive |
| Leukocyte esterase HIGH Positive | Nitrites | HIGH | Positive |
| | Leukocyte esterase | HIGH | Positive |

Abbreviations: LLN=lower limit of normal value provided by the laboratory, ULN=upper limit of normal value provided by the laboratory

All laboratory data will be listed for the Safety Set.

## 7.3 Vital Signs

Descriptive statistics for vital signs (systolic and diastolic blood pressure and pulse rate) and their changes from baseline at each post-baseline visit and at end of study will be presented by treatment group.

Vital sign values will be considered PCI if they meet both the observed value criteria and the change from baseline criteria listed in Table 2. The number and percentage of subjects with PCI post-baseline values will be tabulated by time point and treatment group. The percentages will be calculated relative to the number of subjects with baseline and available assessment at that time point in that treatment group. The numerator is the total number of subjects with at least 1 PCI post-baseline vital sign value at that time point in that treatment group. A supportive listing of subjects with post-baseline PCI values will be provided including the subject number, baseline, and post-baseline PCI values.

Table 2: Criteria for Potentially Clinically Important Vital Signs

| Parameter | Classification | Criteria |
|---|---|---|
| Sitting and Supine | | |
| Systolic BP (mmHg) | LOW and DECREASE | ≤90 and decrease of ≥20 from baseline value |
| Systolic D1 (Illilling) | HIGH and INCREASE | ≥140 and increase of ≥20 from baseline value |
| Diastolic BP | LOW and DECREASE | ≤50 and decrease of ≥15 from baseline value |
| (mmHg) | HIGH and INCREASE | ≥90 and increase of ≥15 from baseline value |
| Pulse rate (bpm) | LOW and DECREASE | ≤45 and decrease of >15 from baseline value |
| Tuise rate (opin) | HIGH and INCREASE | ≥100 and increase of >15 from baseline value |
| Temperature (regardless of method) | LOW | <35°C or <95°F |
| | HIGH | >38.3°C or >100.9°F |
| Respiratory rate | LOW | <10 |
| (breaths/min) | HIGH | >25 |

Abbreviations: BP=blood pressure, bpm=beats per minute.

All vital signs data will be listed for the Safety Set.

## 7.4 Electrocardiogram (ECG)

Descriptive statistics for ECG variables (heart rate, PR, RR, QRS, QT, and QTc intervals) and their changes from baseline at each time point will be presented by treatment group. QTc interval will be calculated using both Bazett (QTcB=QT/(RR)<sup>1/2</sup>) and Fridericia (QTcF=QT/(RR)<sup>1/3</sup>) corrections; and if RR is not available, it will be replaced with 60/(heart rate) in the correction formula. The ECG interpretation at each time point will be summarized by treatment group. A shift table from baseline to each time point for qualitative ECG results will be presented by treatment group.

Electrocardiogram variable values will be considered PCI if they meet or exceed the upper limit values listed in Table 3. The number and percentage of subjects with post-baseline PCI values will be tabulated by treatment and time point. The percentages will be calculated relative to the number of subjects with available non-PCI baseline and available assessment at that time point in that treatment group. The numerator is the total number of subjects with at least 1 PCI post-baseline ECG value at that time point in that treatment group. A listing of all subjects with post-baseline PCI value will be provided including the subject number, baseline, and post-baseline PCI values.

Table 3: Criteria for Potentially Clinically Important ECG Values

| Parameter | Classification | Criteria |
|---|---|---|
| Overall evaluation | ABNORMAL | Overall evaluation is ABNORMAL |
| Rhythm | NON-SINUS | Rhythm is not SINUS |
| Kilytiiii | RHYTHM | Kilytiiii is not siivos |
| Heart rate (bpm) | LOW and DECREASE | ≤45 and decrease of >15 from baseline value |
| Treatt rate (opin) | HIGH and INCREASE | ≥100 and increase of >15 from baseline value |
| PR interval (msec) | HIGH and INCREASE | ≥200 and increase of ≥20 from baseline value |
| QRS interval (msec) | HIGH | ≥120 |
| QTc interval (men) | HIGH | >430 and increase from baseline value >30 |
| (msec)* | mon | > 450 and merease from baseline value > 50 |
| QTc interval (women) | HIGH | >450 and increase from baseline value >30 |
| (msec)* | mon | > 450 and merease from baseline value > 50 |

Abbreviations: bpm=beats per minute; OTc=OT interval corrected.

#### 7.5 Other Safety Data

No other safety assessments/variables are planned for this study.

#### 8. PHARMACOKINETIC ANALYSIS

#### 8.1 Drug Concentration

Blood samples will be drawn from each subject during this study for the determination of plasma concentration of anagrelide, 3-hydroxy-anagrelide, and RL603. Serial blood samples will be collected on Day 1 and Day 8 for PK analysis at predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 8, and 12 hours after administration of the investigational product. Plasma concentrations of anagrelide and its metabolites will be measured using a validated analytical method.

Blood samples will be drawn from each subject during this study for the determination of plasma concentration of omeprazole. Omeprazole PK sample collections on Days 6 and

<sup>\*</sup>Values noted refer to both Bazett's (QTcB) and Fridericia's (QTcF) formula

Day 7 will be taken at pre-dose only. Serial blood samples will be collected on treatment on Day 8 for PK analysis at predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 8, 12, and 24 hours after administration of the investigational product. Plasma concentrations of omeprazole will be measured using a validated analytical method.

# 8.2 Handling Below Limit of Quantitation Values

The following procedures will be used for plasma concentrations of anagrelide and its metabolites and omegrazole data below the lower limit of quantification (LLOQ):

- Samples that are below limit of quantification (BLQ) are reported as <LLOQ on the data listings, where LLOQ is replaced by the actual value for LLOQ for specific PK assay.
- Samples that are BLQ are treated as zero in the calculation of summary statistics (eg, mean, SD, etc.) for the plasma concentrations at individual time points. Geometric mean will be set to missing where zero values exist.
- Mean concentrations are reported as zero if all values are BLQ or zero, and no
  other descriptive statistics are reported. If the calculated mean (± SD)
  concentration is less than the LLOQ, the value will be reported as calculated. The
  mean values derived using these conventions will be used to create the mean
  plasma concentration versus time plots.
- For calculation of area under the curve (AUC), BLQ values are set equal to zero in the dataset loaded into Phoenix<sup>®</sup> WinNonlin<sup>®</sup> (Certara USA, Inc, Princeton, NJ) for PK analysis. WinNonlin<sup>®</sup> uses the zero values that occur before the first time point with a concentration greater than LLOQ. All BLQ values following the first measurable concentration will be set to "missing" in the dataset loaded into WinNonlin<sup>®</sup>.
- Missing values will not be imputed.

#### **8.3** Pharmacokinetic Parameters

Pharmacokinetic parameters will be determined on Day 1 and Day 8 for anagrelide and its metabolites and on Day 8 for omeprazole from the individual plasma concentration versus actual time data. Pharmacokinetic parameters will be estimated by non-compartmental analysis, as deemed appropriate, using Phoenix WinNonlin (Certara USA, Inc., Princeton, NJ) Version 8.0 or higher and all calculations will be based on the actual time since dose.

The PK parameters for anagrelide, 3-hydroxy-anagrelide and RL603 with and without omeprazole administration on Day 1 and Day 8, and PK parameters for omeprazole (and its metabolite) will include, but may not be limited to:

Shire

08 May 2019


| Parameter | Description |
|---|---|
| AUC <sub>0-∞</sub> | Area under the curve extrapolated to infinity, calculated using the observed value of the last non-zero concentration, calculated using the linear up/log down trapezoidal rule (anagrelide and metabolites) |
| AUC <sub>0-t</sub> | Area under the curve from time 0 to the last time point of sample collection, calculated using the linear up/ log down trapezoidal rule (anagrelide and metabolites) |
| AUC <sub>0-tau</sub> | Area under the curve from time 0 to the end of the dosing interval (24 hours post dose), calculated using the linear up/log down trapezoidal rule (omeprazole only) |
| C <sub>max</sub> | Maximum concentration |
| Cmin | Minimum concentration observed over the dosing interval (omeprazole only) |
| Ctrough | Plasma concentration observed at the end of a dosing interval (collected before the next administration [predose concentration at Day 6, Day 7 and Day 8]) (omeprazole only) |
| t <sub>max</sub> | Time of maximum observed concentration sampled during a dosing interval |
| t½ | Terminal half-life, calculated as $ln(2)/\lambda_z$ |
| CL/F | Total body clearance, calculated as: Dose/AUC₀-∞ (anagrelide only) and Dose/AUC₀-tau (omeprazole only) |
| V <sub>z</sub> /F | Volume of distribution associated with the terminal slope following extravascular administration, calculated as: $CL/F / \lambda_z$ (anagrelide and omeprazole only) |
| MRAUC | Metabolite ratio (anagrelide metabolites only), calculated as: AUC₀-∞ (metabolite) / AUC₀-∞ (parent); molecular weight adjustment needed for metabolites. |
| MRC <sub>max</sub> | Metabolite ratio (anagrelide metabolites only), calculated as: C <sub>max</sub> (metabolite) / C <sub>max</sub> (parent); molecular weight adjustment needed for metabolites. |

The primary PK parameters will include the  $C_{max}$ ,  $AUC_{0-t}$ , and  $AUC_{0-\infty}$  for an agrelide and its metabolites, 3-OH-an agrelide (BCH24426) (active) and RL603 (inactive).

# 8.4 Statistical Analysis of Pharmacokinetic Data

Individual anagrelide, 3-hydroxy-anagrelide, RL603, and omeprazole concentrations will be listed by subject, treatment, day, and time and summarized by treatment, day, and time based on the PK Set.

08 May 2019

The following descriptive statistics of plasma concentration summary will be provided: number of subjects, arithmetic mean, geometric mean, SD, arithmetic CV%, geometric CV%, 25th Percentile (Q1), 75<sup>th</sup> Percentile (Q3), median, minimum, and maximum.

The mean and individual plasma anagrelide, 3-hydroxy-anagrelide, and RL603, and omeprazole concentrations versus time profiles by treatment will be presented in figures on both linear and semi-logarithmic scales. Mean (±SD) and individual anagrelide, 3-hydroxy-anagrelide, RL603, and omeprazole plasma concentrations versus time profiles will be presented using nominal time based on the PK Set.

As well as being summarized and presented graphically for all subjects combined, anagrelide, 3-hydroxy-anagrelide, and RL603 concentrations will also be summarized and presented graphically by CYP2C19 metabolizer status (EM and IM/PM). Refer to Section 5.2 for CYP2C19 metabolizer status criteria.

Individual anagrelide, 3-hydroxy-anagrelide, RL603, and omeprazole PK parameters will be listed by subject, treatment, and day, and summarized by treatment and day based on the PK Set with the following descriptive statistics: n, arithmetic mean, arithmetic SD, 95% CI of the mean, CV%, median, Q1, Q3, minimum, maximum, geometric mean, 95% CI of the geometric mean, and geometric CV%.

As well as being performed for all subjects combined, anagrelide, 3-hydroxy-anagrelide, and RL603 parameters will also be analyzed by CYP2C19 metabolizer status (EM and IM/PM).

A linear mixed model using a 2-factor analysis of variance (ANOVA) for a single-sequence crossover design with fixed factors for treatment and subject will be used to compare the log-transformed PK parameters between the 2 treatments (anagrelide with omeprazole versus anagrelide alone). The magnitude of the effect of omeprazole on the PK profile of anagrelide and its metabolites will be evaluated by the point estimate and ninety percent (90%) CIs for the treatment difference on the log-transformed parameters back-calculated to the original scale for the comparisons of C<sub>max</sub>, AUC₀-t, and AUC₀-∞. The geometric mean ratios of the PK parameters comparing anagrelide with omeprazole to anagrelide alone and the corresponding 90% CIs will be calculated for (1) all subjects, (2) EMs, and (3) IMs/PMs.

#### 9. OTHER ANALYSES

No other analyses are planned for this study.

#### 10. INTERIM ANALYSIS/ DATA MONITORING COMMITTEE

There is no planned interim analysis or Data Monitoring Committee in this study.

#### 11. DATA HANDLING CONVENTIONS

#### 11.1 General Data Reporting Conventions

Continuous variables will be summarized using the following descriptive statistics: number of subjects, mean, median, standard deviation, Q1, Q3, minimum, maximum. Categorical and count variables will be summarized by the number of subjects and the percent of subjects in each category.

See Shire TFL Standards for rules on the number of decimal places to present data and *p*-values.

#### 11.2 Definition of Baseline

Baseline for all safety analyses is defined as the last observed value for the safety assessment prior to taking the first dose of investigational product on Day 1 (based on dates or date/times).

## 11.3 Repeated or Unscheduled Assessments of Safety Parameters

If a subject has repeated assessments before the start of investigational product, then the results from the final assessment made prior to the start of investigational product will be used as baseline. If end of study assessments are repeated or unscheduled, the last post-baseline assessment will be used as the end of study assessment for generating descriptive statistics. However, all post-baseline assessments will be used for PCI value determination and all assessments will be presented in the data listings.

#### 11.4 Handling of Missing, Unused, and Spurious Data

# 11.4.1 Missing Date Information for Prior or Concomitant Medications (Therapies/Procedures)

For prior or concomitant medications, incomplete (ie, partially missing) start date and/or stop date will be imputed. When the start date and the stop date are both incomplete for a subject, impute the start date first.

otocol Number: SPD422-113 08 May 2019

#### 11.4.1.1 Incomplete Start Date

The following rules will be applied to impute the missing numerical fields. If the stop date is complete and the imputed start date is after the stop date, then the start date will be imputed using the stop date.

## 11.4.1.1.1 Missing Day and Month

- If the year of the incomplete start date is the same as the year of the date of the first dose of investigational product, then the day and month of the date of the first dose of investigational product will be assigned to the missing fields.
- If the year of the incomplete start date is before the year of the date of the first dose of investigational product, then December 31 will be assigned to the missing fields.
- If the year of the incomplete start date is after the year of the date of the first dose of investigational product, then 01 January will be assigned to the missing fields.

# 11.4.1.1.2 Missing Month Only

• The day will be treated as missing and both month and day will be replaced according to the above procedure.

# **11.4.1.1.3 Missing Day Only**

- If the month and year of the incomplete start date are the same as the month and year of the date of the first dose of investigational product, then the day of the date of the first dose of investigational product will be assigned to the missing day
- If either the year is before the year of the date of the first dose of investigational product or if both years are the same, but the month is before the month of the date of the first dose of investigational product, then the last day of the month will be assigned to the missing day
- If either the year is after the year of the date of the first dose of investigational product or if both years are the same, but the month is after the month of the date of the first dose of investigational product, then the first day of the month will be assigned to the missing day.

# 11.4.1.2 Incomplete Stop Date

The following rules will be applied to impute the missing numerical fields.

#### 11.4.1.2.1 Missing Day and Month

- If the year of the incomplete stop date is the same as the year as of the date of the last dose of investigational product, then the day and month of the date of the last dose of investigational product will be assigned to the missing fields.
- If the year of the incomplete stop date is before the year of the date of the last dose of investigational product, then 31 December will be assigned to the missing fields.

• If the year of the incomplete stop date is after the year of the date of the last dose of investigational product, then 01 January will be assigned to the missing fields.

# 11.4.1.2.2 Missing Month Only

• The day will be treated as missing and both month and day will be replaced according to the above procedure.

# **11.4.1.2.3 Missing Day Only**

- If the month and year of the incomplete stop date are the same as the month and year of the date of the last dose of investigational product, then the day of the date of the last dose of investigational product will be assigned to the missing day
- If either the year is before the year of the date of the last dose of investigational product or if both years are the same, but the month is before the month of the date of the last dose of investigational product, then the last day of the month will be assigned to the missing day
- If either the year is after the year of the last dose of investigational product or if both years are the same, but the month is after the month of the date of the last dose of investigational product, then the first day of the month will be assigned to the missing day.

# 11.4.2 Missing Date Information for Adverse Events

For AEs with partial start dates, non-missing date parts will be used to determine if the AE is treatment-emergent or not. If a determination cannot be made using the non-missing date parts as to when the AE occurred relative to study drug administration, eg, AE start year and month are the same as the year and month of the first dose of investigational product, then the AE will be classified as treatment-emergent.

To facilitate categorization of AEs as treatment-emergent, imputation of dates can be used. For AEs, the default is to only impute incomplete (ie, partially missing) start dates. Incomplete stop dates may also be imputed when calculation of the duration of an AE is required per the protocol. If imputation of an incomplete stop date is required, and both the start date and the stop date are incomplete for a subject, impute the start date first.

#### 11.4.2.1 Incomplete Start Date

Follow the same rules as in Section 11.4.1.1.

#### 11.4.2.2 Incomplete Stop Date

Follow the same rules as in Section 11.4.1.2.

# 11.4.3 Missing Severity Assessment for Adverse Events

If severity is missing for an AE starting prior to the date of the first dose of investigational product, then a severity of "Mild" will be assigned. If the severity is missing for an AE starting on or after the date of the first dose of investigational product, then a severity of "Severe" will be assigned. The imputed values for severity assessment will be used for incidence summaries, while both the actual and the imputed values will be used in data listings.

# 11.4.4 Missing Relationship to Investigational Product for Adverse Events

If the relationship to investigational product is missing for an AE starting on or after the date of the first dose of investigational product, a causality of "Related" will be assigned. The imputed values for relationship to investigational product will be used for incidence summaries, while both the actual and the imputed values will be presented in data listings.

# 11.4.5 Character Values of Clinical Laboratory Variables

If the reported value of a clinical laboratory variable cannot be used in a statistical analysis due to, for example, that a character string is reported for a numerical variable. The appropriately determined coded value will be used in the statistical analysis. However, the actual values as reported in the database will be presented in data listings.

#### 12. ANALYSIS SOFTWARE

Statistical analyses will be performed using Version 9.4 (or newer) of SAS® on a suitably qualified environment.

Phoenix WinNonlin (Certara USA, Inc., Princeton, NJ) Version 8.0 (or higher) will be used for calculation of PK parameters.

#### 13. CHANGES TO ANALYSIS SPECIFIED IN PROTOCOL

Not applicable.

Shire 

Shire Statistical Analysis Plan v1.0 Protocol Number: SPD422-113

08 May 2019

# 14. REFERENCES

Not applicable.

# 15. APPENDICES

# 15.1 Schedule of Activities

Table 4: Schedule of Assessments

| | Screening<br>Period | | Treatment<br>Period | | | | | | | | Early<br>Termination <sup>a</sup> | Follow Up<br>Phone | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day -28 to<br>Day -2 | Day -1 | Day 1 | Day 2 | Day 3 | Day 4 | Day 5 | Day 6 | Day 7 | Day 8 | Day 9 | | Contact 7±2<br>days <sup>b</sup> |
| Informed Consent | X | | | | | | | | | | | | |
| In-Patient <sup>c</sup> | | X | X | X | X | X | X | X | X | X | X | | |
| Inclusion/Exclusion Criteria | X | X | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | |
| Medical & Medication History | X | | | | | | | | | | | | |
| Physical Examination | X | X | X | | | | | | | | X | X | |
| Height, weight and calculate BMId | | | | | | | | | | | | | |
| Vital Signs (blood pressure and pulse) <sup>e</sup> | X | X | X | | | | | | | X | X | X | |
| 12-lead ECG e | X | X | X | | | | | | | X | X | X | |
| Drugs of abuse and alcohol screen | X | X | | | | | | | | | | | |
| Urine cotinine | X | X | | | | | | | | | | | |
| HIV, HBsAg, and HCV screen | X | | | | | | | | | | | | |
| Serum Pregnancy (all females) | X | X | | | | | | | | | X | X | |
| Biochemistry, hematology, and urinalysis | X | X | X | | | | | | | X | X | X | |
| TSH and T4 | X | | | | | | | | | | | | |
| Omeprazole PK Sample<br>Collection <sup>f</sup> | | | | | | | | X f | X f | X | X | | |
| Anagrelide PK Sample Collection | | | X | | | | | | | X | | | |
| Administration of omeprazole <sup>g</sup> | | | | X | X | X | X | X | X | Xi | | | |
| Administration of anagrelide h, i | | | X i | | | | | | | X i | | | |
| Concomitant Medications | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Adverse events/serious adverse events | X | X | X | X | X | X | X | X | X | X | X | X | X |

BMI=body mass index; ECG=electrocardiogram; HIV=human immunodeficiency virus, HBsAG=hepatitis B surface antigen, HCV=hepatitis C virus; TSH=thyroid stimulating hormone, T4=thyroxine, PK=pharmacokinetic

- <sup>a</sup> An attempt to perform the early termination assessments and procedures will be made for any subject who withdraws or is removed from the study.
- <sup>b</sup> A follow up telephone contact (or in-person follow-up contact at the investigator's discretion) will take place 7±2 days following the subject's last dose of anagrelide.
- <sup>c</sup> Subjects will remain in-patient at the Clinical Research Center starting on Day -1 until discharged following the 24-hour post dose PK sample and safety assessments on the morning of Day 9
- <sup>d</sup> Height to be measured without shoes and weight to be taken in light clothes
- <sup>e</sup> Subjects should be resting in a supine position for at least 5 minutes prior to collecting vital signs and ECGs. Vital sign assessments during the screening visit only include blood pressure, pulse, respiratory rate and temperature.
- <sup>f</sup> Omeprazole PK sample collections on Days 6 and Day 7 are to be taken at pre-dose only.
- <sup>g</sup> Omeprazole is to be administered prior to breakfast.
- h Anagrelide should be taken by the subject at 8:00 am. If more than 1 subject is receiving anagrelide on the same day, the dosing interval between subjects may be a stagger of 3 minutes between dose administrations.
- <sup>1</sup> Subjects are required to fast for approximately 10 hours prior to and until 4 hours post dose (after PK and safety assessments) on Days 1 and 8.

Table 5: Schedule of Assessments – Detail of Treatment Period Day 1

| Study Procedure/Relative to IP Administration | Administration<br>of<br>Anagrelide <sup>a</sup> | Anagrelide<br>PK Sample<br>Collection | Physical<br>Examination | Vital Signs <sup>b</sup><br>(BP and<br>pulse) | 12-lead<br>ECG <sup>b</sup> | Biochemistry,<br>hematology,<br>and urinalysis | Concomitant<br>Medications | Adverse<br>Events/Serious<br>Adverse Events |
|---|---|---|---|---|---|---|---|---|
| Pre-dose <sup>c</sup> | | X | | X | X | X | X | X |
| 0 | X <sup>d</sup> | | | | | | X | X |
| 0.5 hours | | X | | | | | X | X |
| 1 hour | | X | | X | | | X | X |
| 1.5 hours | | X | | | | | X | X |
| 2 hours | | X | | X | | | X | X |
| 2.5 hours | | X | | | | | X | X |
| 3 hours | | X | | | | | X | X |
| 4 hours | | X | | X | | | X | X |
| 8 hours | | X | | X | | | X | X |
| 12 hours | | X | X | X | X | X | X | X |

ECG=electrocardiogram; PK=pharmacokinetic; IP=investigation product

<sup>&</sup>lt;sup>a</sup> The subjects should be administered anagrelide starting at 8:00 am.

<sup>&</sup>lt;sup>b</sup> Subjects should be resting in a supine position for at least 5 minutes prior to collecting vital signs and ECGs.

<sup>&</sup>lt;sup>c</sup> Pre-dose assessments should be performed within 30 minutes prior to dose.

<sup>&</sup>lt;sup>d</sup> Subjects are required to fast for approximately 10 hours prior to and until 4 hours post-dose (after PK and safety assessments) on Day 1 and 8.

Table 6: Schedule of Assessments – Detail of Treatment Period Day 8

| Study Procedure/Relative to IP Administration | Administration<br>of Anagrelide<br>&<br>Omeprazole <sup>a</sup> | Anagrelide<br>PK Sample<br>Collection | Omeprazole<br>PK Sample<br>Collection | Physical<br>Examination | Vital Signs <sup>b</sup><br>(BP and pulse) | 12-lead<br>ECG <sup>b</sup> | Biochemistry,<br>hematology,<br>and urinalysis | Concomitant<br>Medications | Adverse<br>Events/Serious<br>Adverse<br>Events |
|---|---|---|---|---|---|---|---|---|---|
| Pre-dose <sup>c</sup> | | X | X | | X | X | X | X | X |
| 0 | X <sup>d</sup> | | | | | | | X | X |
| 0.5 hours | | X | X | | | | | X | X |
| 1 hour | | X | X | | X | | | X | X |
| 1.5 hours | | X | X | | | | | X | X |
| 2 hours | | X | X | | X | | | X | X |
| 2.5 hours | | X | X | | | | | X | X |
| 3 hours | | X | X | | | | | X | X |
| 4 hours | | X | X | | X | | | X | X |
| 8 hours | | X | X | | X | | | X | X |
| 12 hours | | X | X | | X | X | | X | X |
| 24 hours | | | X | X | X | X | X | X | X |

ECG=electrocardiogram; PK=pharmacokinetic; IP=investigation product

<sup>&</sup>lt;sup>a</sup> The subjects should be administered anagrelide and omeprazole concurrently starting at 8:00 am.

<sup>&</sup>lt;sup>b</sup> Subjects should be resting in a supine position for at least 5 minutes prior to collecting vital signs and ECGs.

<sup>&</sup>lt;sup>c</sup> Pre-dose assessments should be performed within 30 minutes prior to dose.

<sup>&</sup>lt;sup>d</sup> Subjects are required to fast for approximately 10 hours prior to and until 4 hours post-dose (after PK and safety assessments) on Days 1 and Day 8.